CLINICAL TRIAL: NCT04126954
Title: Multicentric Retrospective Study on the Use of Cinacalcet in an Off-label Phosphocalcic Context
Brief Title: Study on the Use of Cinacalcet in Phosphocalcic Context.
Acronym: CALCI-CINA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2019_CALCI-CINA
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Hyperparathyroidism, Secondary; Hyperparathyroidism, Primary
Keywords: Hyperparathyroidism; pathology phosphocalcic
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Hyperparathyroidism, Primary; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cinacalcet: Patients with primary or secondary hyperPTH resulting from phosphocalcic pathology treated by cinacalcet
  Interventions: Other: Serum PTH concentrations results

INTERVENTIONS:
Other: Serum PTH concentrations results — To compare serum PTH concentrations results in patients with primary or secondary hyperPTH resulting from phosphocalcic pathology before and three months after initiation of cinacalcet therapy.

SUMMARY:
Currently, the indications used for MA (Marketing Authorization) Cinacalcet in France are hyperparathyroidism (hyperPTH) in adults, whether primary (for patients in whom parathyroidectomy is theoretically indicated but in whom it is contraindicated or not is not clinically appropriate) or secondary to a chronic kidney disease, and parathyroid carcinomas.

In pediatric patients, data on its use are restricted due to its recent marketing authorization (2017) and limited to dialysis patients suffering from secondary hyperPTH.

Nevertheless, some patients with phosphocalcic pathologies without renal insufficiency must be treated off-label by cinacalcet in the presence of severe hyperPTH, without any other chronic treatment available to date.

The objective of this study is therefore to evaluate the use in France of cinacalcet in phosphocalcic pathologies without renal insufficiency, in order to obtain efficacy and safety data in order to improve our knowledge on the management of these orphan diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with phosphocalcic pathology without end-stage renal failure
* Patients followed in one of the hospitals of the centers of reference and competence of the diseases of the metabolism of calcium and phosphate
* For children under 18: patient and parent (s) / parent having been informed of the study and having expressed their on-opposition
* For adults: patient / legal guardian of the patient under guardianship having been informed of the study and expressing his or her non opposition

Exclusion Criteria:

* Patient suffering from parathyroid cancer,
* Patient suffering from primary hyperPTH in whom parathyroidectomy would theoretically be indicated but contraindicated or clinically inappropriate,
* Patient suffering from hyperPTH secondary to end-stage renal failure
* No social security support

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with phosphocalcic diseases suffering from hyperPTH without end-stage renal failure.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Serum PTH concentration | 3 months after treatment initiation

SECONDARY OUTCOMES:
Serum PTH concentration | 1 month after treatment initiation
Serum PTH concentration | 6 months after treatment initiation
Serum PTH concentration | 12 months after treatment initiation
Serum PTH concentration | 3 years after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Justine BACCHETTA, MD, Principal Investigator — Service de Néphrologie, Rhumatologie et Dermatologie Pédiatriques
Locations (10):
- France (10):
  - Endocrinologie Diabète et Maladies Métaboliques - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Service de Néphrologie Pédiatrique -Hôpital Jeanne de Flandre, Lille
  - Service d'Endocrinologie Pédiatrique - Hôpital de la mère et de l'Enfant, Limoges
  - Pole Femme Mère Enfant - Pédiatrie spécialisée - Centre Hospitalier Universitaire, Montpellier
  - Service de Néphrologie pédiatrique - Clinique Médicale Pédiatrique, Nantes
  - Service d'endocrinologie et Diabétologie Pédiatrique-Hôpital Robert Debré, Paris
  - Service de Diabétologie et endocrinologie pédiatriques - Centre Hospitalier Universitaire, Reims
  - Pôle Néphrologie-Urologie-Diabétologie-Endocrinologie, Strasbourg
  - Service d'Endocrinologie, Maladies Osseuses, Gynécologie, Génétique, Toulouse
  - Unité Endocrinologie, Nutrition, Diabétologie -Hôpital Bretonneau, Tours